CLINICAL TRIAL: NCT01078792
Title: Prognostic Value of Prothrombin Fragments 1+2 for Pulmonary Embolism Incidence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Marinella Beckerman, Hillel Yaffe Medical Center
Other Study IDs: 0001-10
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Disease Exacerbation; Pulmonary Embolism; Prothrombin Fragments
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease Progression; Pulmonary Embolism | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD exacerbation: Patients admitted to hospital with COPD exacerbation
  Interventions: Other: CT pulmonary angio, blood tests

INTERVENTIONS:
Other: CT pulmonary angio, blood tests

SUMMARY:
To determine the possible association of prothrombin fragments 1+2 elevation with incidents of pulmonary embolism in patients with COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* COPD exacerbation
* Able to give informed consent
* Able to perform spirometry

Exclusion Criteria:

* Known malignancy
* Known hypercoagulable state
* Receiving anticoagulant treatment
* Pregnancy
* Renal failure
* Allergy to Iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital due to COPD exacerbation
Sampling Method: Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel